CLINICAL TRIAL: NCT03044002
Title: BIOTRONIK 4French for AMBulatory Peripheral Intervention. A Multicenter, Controlled Trial Comparing 4French Versus 6French Femoral Access for Endovascular Treatment of Lower-extremity Peripheral Artery Disease in an Ambulatory Setting: BIO4AMB
Brief Title: BIOTRONIK 4French for AMBulatory Peripheral Intervention
Acronym: BIO4AMB
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1602
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Artery Disease; Access Site Complication; Outpatient Treatment
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- 4French Intervention: Patient with infrainguinal Peripheral Artery Disease (PAD), requiring endovascular treatment
  Interventions: Device: Biotronik 4 French Portfolio
- 6French Intervention: Patient with infrainguinal Peripheral Artery Disease (PAD), requiring endovascular treatment
  Interventions: Device: 6 French Portfolio

INTERVENTIONS:
Device: Biotronik 4 French Portfolio — Ambulatory intervention by femoral access for endovascular treatment of lower-extremity peripheral artery disease
  Groups: 4French Intervention
Device: 6 French Portfolio — Ambulatory intervention by femoral access for endovascular treatment of lower-extremity peripheral artery disease
  Groups: 6French Intervention

SUMMARY:
BIOTRONIK 4French for AMBulatory peripheral intervention. A multicenter, controlled trial comparing 4French versus 6French femoral access for endovascular treatment of lower-extremity peripheral artery disease in an ambulatory setting: BIO4AMB

DETAILED DESCRIPTION:
Controlled, multicenter, non-inferiority trial to compare the rate of access site complications (ASC) in 4French (4F) vs. 6French (6F) femoral access endovascular interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* Ability to walk
* Subject must be willing to sign patient Informed Consent (PIC)
* Patient with infrainguinal arteries lesion(s) suitable to be treated during an ambulatory endovascular intervention

Exclusion Criteria:

* No possibility of an ambulatory management
* Physical fitness classified as ASA ≥ 4 (American Society of Anaesthesiologists)
* Coagulation disorders
* Acute ischemia
* Less than 1month live expectancy
* Pregnant or breast feeding females or females who intend to become pregnant during the time of the study (pregnancy test required for all women with child bearing potential)
* Subject currently enrolled in other medical or drug study and has not reached the primary outcome measures
* Patient contraindicated for antiplatelet therapy, anticoagulants and antithrombotics
* Other access than common femoral
* Home alone the first night

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with infrainguinal Peripheral Artery Disease (PAD), requiring endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Peri- and post-procedural access site complications (including homeostasis strategy failure; post-procedural defined as within 30 days post-intervention) | up to 30 days post procedure
  Access site complications are defined as a composite of:
  * Groin hematoma (larger than 5 cm in diameter, visible by sonography, and hemoglobin decrease <3 g/dL)
  * Pseudoaneurysm
  * Groin as well as retroperitoneal bleeding (defined as requiring acute intervention for haemostasis, need for blood transfusions, or haemoglobin decrease >3 g/dL)
  * AV fistula (visible by shunting in colour coded sonography between the common femoral artery and vein)
  * Arterial dissections at access site (visible with fluoroscopy or sonography as a membrane causing stenosis in the vessel lumen)
  * Thrombosis
  * VCD related ASCs

CONTACTS AND LOCATIONS:
Overall Officials: PD Dott. med. Jos van den Berg, Principal Investigator — Ospedale Regionale di Lugano - Sezione Civico; a.o. Univ. Prof. Dr. Marianne Brodmann, Principal Investigator — Substitute Head of the Clinical Division of Angiology, Department of Internal Medicine
Locations (5):
- Medizinische Universitaet Graz, Graz, Austria
- A.Z.Sint-Blasius, Dendermonde, Belgium
- France (2):
  - CHU du Bocage, Dijon
  - Clinique Saint Joseph, Trélazé
- Osepedale Regionale di Lugano, Lugano, Switzerland